CLINICAL TRIAL: NCT06902935
Title: Establishment and Clinical Application of Breast Cancer Risk Prediction Model Based on Traditional Chinese Medicine Four Diagnostic Instruments and Ultrasound
Status: Not yet recruiting | Type: Observational
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Sun Mengwei, Establishment and Clinical Application of Breast Cancer Risk Prediction Model Based on Traditional Chinese Medicine Four Diagnostic Instruments and Ultrasound, Taizhou Hospital
Other Study IDs: 2025L-02-012
Record Dates: First submitted 2025-02-16; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group: The patients included in the group are those whose pathological results of breast masses are malignant.
  Interventions: Diagnostic Test: Diagnosis of Breast Cancer by Traditional Chinese Medicine Four Examinations
- Control group: The patients included in this group are those whose pathological results of breast masses are benign.
  Interventions: Diagnostic Test: Ultrasound diagnosis of breast cancer

INTERVENTIONS:
Diagnostic Test: Diagnosis of Breast Cancer by Traditional Chinese Medicine Four Examinations — The Daosheng TCM Four-Diagnostic Instrument (DS01-A) comprehensively collects patients' TCM four-diagnostic information, covering tongue (e.g., overall color, coating color/thickness/greasiness, tooth marks, etc.), pulse (e.g., position, force, rhythm, etc.), face (e.g., overall color, luster, lip color/dryness, etc.) and constitution scores (quantifying 9 constitutions via the TCM Constitution Classification Table).
  Groups: Case group
Diagnostic Test: Ultrasound diagnosis of breast cancer — Professional ultrasound physicians use B - ultrasound equipment of the same model to accurately collect detailed parameters of breast masses according to a standardized process. These parameters include shape (oval, round, irregular), orientation (parallel, non - parallel), margin (smooth, non - smooth, with non - smooth including blurred, angular, microlobulated, spiculated, etc.), echo pattern (anechoic, hyperechoic, complex cystic - solid echo, hypoechoic, isoechoic, heterogeneous echo), posterior echo characteristics (no change, enhancement, shadowing, mixed), calcification (microcalcification and coarse calcification within the mass, calcification outside the mass, intraductal), and vascular supply (no blood supply, internal blood supply, marginal blood supply), etc.
  Groups: Control group

SUMMARY:
Construct a breast cancer risk prediction model based on traditional Chinese medicine four diagnostic instruments and B-ultrasound images. Ensure that the key evaluation indicators of the model reach a high level through clinical verification, so as to contribute to accurate clinical diagnosis and treatment decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged between 30 and 75.
2. Patients who have a mass detected by US examination, need to undergo surgery or needle biopsy, and obtain a definite pathological result.
3. Patients who have obtained complete identification results of tongue, pulse, face, and constitution through the traditional Chinese medicine four diagnostic instruments.

Exclusion Criteria:

- 1. Patients with severe heart, liver, or kidney insufficiency, or other serious systemic diseases.

2. Patients with a history of other malignant tumors. 3. Cases with poor - quality B - ultrasound images. 4. Cases with an unclear pathological diagnosis. 5. Patients with obvious lesions on the face, in the oral cavity, or on the tongue that may affect the measurement results.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast masses who come to the clinic for medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-04-26 (Estimated); Primary Completion 2027-04-26 (Estimated); Study Completion 2027-04-26 (Estimated)

PRIMARY OUTCOMES:
Tongue appearance collection (overall tongue color) | through study completion, an average of 1 year
  pale white, pale purple, light red, dark red, dark purple
Tongue appearance collection (overall tongue coating color) | through study completion, an average of 1 year
  white, yellow, no tongue coating
Tongue appearance collection (thickness of the tongue coating) | through study completion, an average of 1 year
  Thin tongue coating, thick tongue coating, scanty tongue coating or no tongue coating
Pulse condition collection (pulse strength) | through study completion, an average of 1 year
  forceful, moderate, weak
Pulse condition collection (pulse rhythm) | through study completion, an average of 1 year
  Regular, rapid intermittent pulse, slow intermittent pulse.
Pulse condition collection (pulse rate) | through study completion, an average of 1 year
  Slow pulse, moderate pulse, normal pulse, rapid pulse, extremely rapid pulse.
Collection of facial appearances (overall facial complexion) | through study completion, an average of 1 year
  Normal facial complexion, white complexion, yellow complexion, red complexion, cyan complexion, black complexion
Collection of facial appearances (overall luster) | through study completion, an average of 1 year
  With luster, without luster
Judgment of Constitution Score | through study completion, an average of 1 year
  Balanced constitution, Qi-deficiency constitution, Yang-deficiency constitution, Yin-deficiency constitution, Phlegm-dampness constitution, Damp-heat constitution, Blood-stasis constitution, Qi-stagnation constitution, Special constitution.

CONTACTS AND LOCATIONS:
Locations (1):
- Taizhou Central Hospital (Affiliated Hospital of Taizhou University), Taizhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided